CLINICAL TRIAL: NCT00458991
Title: Recombinant Human Growth Hormone Therapy and Drug Metabolism
Brief Title: rhGH Therapy on Hepatic Drug Metabolism
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PPRU 10734; U10HD045934-01 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Growth Hormone Deficiency, Dwarfism
Keywords: Recombinant Human Growth Hormone; growth hormone deficiency; short stature; phenotyping
MeSH Terms: conditions — Dwarfism, Pituitary; Dwarfism | interventions — Dextromethorphan; Caffeine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dextromethorphan and Caffeine — All subjects received standard medical therapy with rhGH and at specified times low doses of the pharmacologic "probes" (e.g., caffeine and dextromethorphan) as surrogate markers to determine CYP450 activity. The only direct treatment effect measured was the biological response to rhGH.

SUMMARY:
The purpose of the study is to understand the effect of rhGH therapy on hepatic drug metabolism in children with idiopathic growth hormone deficiency.

DETAILED DESCRIPTION:
Growth Hormone (GH) deficiency is a prominent cause of short stature, affecting approximately 14,000 children in the US. Although a single study has demonstrated reduces CYP1A2 activity following Gh replacement therapy, the effect of GH on the most abundant phase 1 biotransformation pathways (e.g. CYP2D6 and CYP3A4) remain largely uncharacterized. This information gap exists largely due to the lack of sufficiently safe, specific and non-invasive methods appropriate for the longitudinal evaluation of enzyme activity in young children. We can overcome these problems by employing validated phenotyping methods using caffeine, a commonly ingested dietary substance and dextromethorphan, a safe, non-sedating over the counter anti-tussive agent. Application of these methods will permit us to identify, characterize and describe the isoform-specific effects of rhGH on major phase 1 hepatic drug biotransformation pathways, thereby addressing this information gap with minimal risk to children.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 4 to 14 years with a height less than the 5th percentile for age and sex or having a decelerated across two major percentiles (5th, 10th, 25th, 50th, 90th, and 95th) on standard pediatric growth curves, poor growth velocity (less than 5 centimeters/year), radiographic evidence of delayed bone age (i.e. greater than 1 SD below the mean for chronological age) and a documented diagnosis of idiopathic growth hormone deficiency [as determined by failure to raise serum GH concentrations 10 microgram/Liter following provocative testing with two growth hormone secretagogues(e.g. insulin, arginine, or clonidine)].
* All subjects will be prepubertal, as determined by Tanner staging.

Exclusion Criteria:

* Children receiving medications known to induce or inhibit hepatic CYP1A2, NAT-2, XO, CYP2D6 or CYP3A4 activity.
* Subjects with a history of smoking (including exposure to second hand smoke > 8 hours per day) or illicit drug use.
* Subjects with a history of hepatic, renal, cardiac or thyroid disorders. Presence of hepatic, renal, cardiac or thyroid disease will be established based on clinical history and results of recent laboratory tests conducted as part of the routine medical evaluation of children who are being considered for rhGH therapy.
* Children experiencing fever or acute viral illness
* Children who have a history of a hypersensitivity reaction to dextromethorphan or caffeine
* Children who have received prior treatment with rhGH
* Children who are receiving corticosteroids or thyroid hormone

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children recently diagnosed with idiopathic GH deficiency who were candidates for rhGH therapy were eligible for enrollment. All subjects were recruited via informed parental consent and patient assent (for children > 7 years). The anticipated sample size was 12 children.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2001-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Kennedy, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - University of California at San Diego, San Diego, California
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio